CLINICAL TRIAL: NCT02699697
Title: A Prospective Randomized Phase II Study of 1 vs 2 Fractions of Palliative Radiation Therapy for Patients With Symptomatic Bone Metastasis
Brief Title: Palliative Radiation Therapy in Reducing Pain in Patients With Bone Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00037248; NCI-2016-00204 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01416 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm; Metastatic Malignant Neoplasm in the Bone; Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ARM I (palliative radiation therapy) (Experimental): Patients undergo 1 fraction of EBRT over 30 minutes.
  Interventions: Radiation: External Beam Radiation Therapy; Radiation: Palliative Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- ARM II (palliative radiation therapy) (Experimental): Patients undergo 2 fractions of EBRT over 30 minutes. The 2 fractions will be separated by 3-7 days.
  Interventions: Radiation: External Beam Radiation Therapy; Radiation: Palliative Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Radiation: Palliative Radiation Therapy — Undergo EBRT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well palliative radiation therapy works in reducing pain in patients with cancer that has spread from the original (primary) tumor to the bone (bone metastasis). Palliative radiation therapy using external beam radiation therapy may help patients with bone metastasis to relieve symptoms and reduce pain caused by cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether 8 gray (Gy) x 2 fractions results in lower re-treatment rates compared to 8 Gy x 1 fraction.

SECONDARY OBJECTIVES:

I. To determine whether 8 Gy x 2 fractions provides superior pain and narcotic relief compared to 8 Gy x 1 fraction.

II. To determine whether 8 Gy x 2 fractions is associated with improved quality of life compared to 8 Gy x 1 fraction.

III. To determine whether use of a bone strengthening agent is associated with improved pain relief, narcotic relief and re-treatment rates.

IV. To determine if 8 Gy x 2 fractions is associated with increased toxicity. V. To correlate patient satisfaction, perceived stress, and social support with treatment outcomes.

TERTIARY OBJECTIVES:

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo 1 fraction of external beam radiation therapy (EBRT) over 30 minutes.

ARM II: Patients undergo 2 fractions of EBRT over 30 minutes. The 2 fractions will be separated by 3-7 days.

After completion of study treatment, patients are followed up at 30 days and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer, not including multiple myeloma
* Radiographic evidence of bone metastases within 8 weeks of study; the patient must have pain which appears to be related to the radiographically documented metastasis in the opinion of the treating physician, and the decision has been made by the responsible clinician that a course of palliative external beam radiation therapy is appropriate treatment; multiple sites eligible if they can be included in no greater than 3 treatment sites
* Eligible treatment sites are:

  * Weight bearing sites

    * Pelvis (excluding pubis)
    * Femur
    * Sacrum and/or sacroiliac joints
    * Tibia
  * Non-weight bearing sites

    * Up to 5 consecutive cervical, thoracic or lumbar vertebral bodies
    * Lumbosacral spine
    * Up to 3 consecutive ribs
    * Humerus
    * Fibula
    * Radius ± ulna
    * Clavicle
    * Sternum
    * Scapula
    * Pubis If multiple sites are treated, the treatment site is included as weight-bearing if any of the sites include the pelvis, sacrum, femur or tibia
* Pain score of at least 5 on a scale of 0 - 10 within a week of enrollment OR pain score < 5 with >= 60 mg of morphine (or equivalent) per day
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 3
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document
* Negative pregnancy test at study registration
* Changes in systemic chemotherapy, hormonal therapy or the use of bisphosphonates for 4 weeks before and after the delivery of radiotherapy are allowed, but recording and accounting for this in the statistical analysis is required
* Life expectancy of at least 12 weeks as deemed by the treating oncologist
* Patients will be eligible for treatment of multiple osseous sites only if those sites can be included in no more than three treatment sites; for patients with painful metastases that are contiguous but do not fit into the definition of a site listed above, those patients will still be eligible but will be considered to have two treatment sites; for example, a patient with a lesion of T4, T7 and T9 would be eligible but would be considered as two treatment sites since more than five consecutive vertebral bodies would be treated; these lesions could be treated with one field, even though the treatment is coded as two sites

Exclusion Criteria:

* Previous radiotherapy or palliative surgery to the painful site
* Metastases to the skull, hands, feet are not eligible treatment sites
* Spinal cord or cauda equine compression/effacement in vertebral metastases with neurological symptoms other than just pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-05; Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris R Brown, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Control) 8 Gy x 1: Patients undergo 1 fraction of EBRT over 30 minutes.
- Arm B (Treatment) 8 Gy x 2: Patients undergo 2 fractions of EBRT over 30 minutes. The 2 fractions will be separated by 3-7 days.
Period: Overall Study
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Started | 51 | 51
Completed | 19 | 24
Not Completed | 32 | 27
Not completed — Death | 18 | 15
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Refused to follow up | 1 | 1
Not completed — Entered hospice care | 5 | 2
Not completed — Missing reason for discontinuation | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2 | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (14.0) | 64.8 (10.8) | 63.35 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 29 | 30 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 1 | 2
  Ethnicity: Not Hispanic or Latino | 50 | 50 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 40 | 42 | 82
  Race: Black or African American | 9 | 6 | 15
  Race: Asian Indian/Asian | 1 | 1 | 2
  Race: Unable to obtain | 1 | 2 | 3
Currently using bisphosphonates/ Denosumab? [Count of Participants; unit: Participants] | 10 | 4 | 14
Any prior cancer therapy [Count of Participants; unit: Participants] | 32 | 24 | 56
History of weight loss? [Count of Participants; unit: Participants] | 18 | 16 | 34
Medical History [Count of Participants; unit: Participants]
  Myocardial infarction | 3 | 1 | 4
  Congestive heart failure | 2 | 2 | 4
  Peripheral vascular disease | 2 | 0 | 2
  Cerebrovascular disease | 6 | 5 | 11
  Dementia | 0 | 1 | 1
  Chronic pulmonary disease | 3 | 8 | 11
  Connective tissue disease | 0 | 2 | 2
  Peptic ulcer disease | 2 | 2 | 4
  Liver disease | 0 | 1 | 1
  Diabetes | 5 | 12 | 17
  Hemiplegia | 1 | 1 | 2
  Other cancer | 14 | 15 | 29
  AIDS | 0 | 0 | 0
  Other sites of metastases | 37 | 35 | 72
  Brain | 9 | 8 | 17
  Liver | 13 | 12 | 25
ECOG Performance Status [Count of Participants; unit: Participants] — Score 0 - Fully active, able to carry on all pre-disease performance without restriction.
  Score 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Score 2 - Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Score 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  Participants
    0-1 | 31 | 34 | 65
    2-3 | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Re-Treatment Rates - Arm 1 (8 Gy x 1) vs. Arm 2 (8 Gy x 2)
Description: The primary analysis will use a one-sided Z-test for proportions to test the null hypothesis.
Time Frame: Up to 6 months post-treatment
Population: Analysis was performed with death as a competing risk.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 45 | 46
Participants
  Retreatment | 3 | 3
  Death | 19 | 17
Statistical Analysis 1: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Test type: Superiority; p = 0.8325, t-test, 2 sided; Hazard Ratio (HR) = 0.869

2. Secondary Outcome: Change in Pain Intensity Assessed Using the Numerical Rating Pain Scale NRPS - Continuous Scale
Description: Measured on a continuous scale and will be compared between groups using 2-sample t-tests. Pain, on a 0-10 scale, and narcotic use, in daily oral morphine equivalents, by treatment arm assessed at 3 and 6 months post-treatment completion.
Time Frame: At 3 months and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 19 | 24
score on a scale
  Continuous scale - 3 months | 4.4 (3.7) | 3.8 (3.1)
  Continuous scale - 6 months | 4.2 (3.6) | 4.4 (3.0)
Statistical Analysis 1: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Continuous pain scale p-value at 3 months; Test type: Superiority; p = 0.5593, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Continuous pain scale p-value at 6 months; Test type: Superiority; p = 0.8133, t-test, 2 sided

3. Secondary Outcome: Change in Narcotic Use Assessed Using the Numerical Rating Pain Scale NRPS - Narcotic Use
Description: Measured on a continuous scale and will be compared between groups using 2-sample t-tests. Pain, on a 0-10 scale, and narcotic use, in daily oral morphine equivalents, by treatment arm assessed at 3 and 6 months post-treatment completion.
  The variable for pain response is categorical rather than continuous and will be compared between groups using a Fisher's exact test. The rating pain scale is from 0-10, with 0 being no pain, 8-10 worst possible pain.
Time Frame: At 3 months and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: MME per day
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 19 | 24
MME per day
  Narcotic use in daily morphine equivalents - 3 months | 6 (18.2) | 9 (29.0)
  Narcotic use in daily morphine equivalents - 6 months | 5 (7.3) | 6 (5.0)
Statistical Analysis 1: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Narcotic use at 3 months; Test type: Superiority; p = 0.3058, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Narcotic use at 6 months; Test type: Superiority; p = 0.5337, t-test, 2 sided

4. Secondary Outcome: Change in Quality of Life Measured Using the Quality of Life Questionnaire (QLQ) Core(C)15-palliative (PAL)
Description: Analyses will be performed that examine whether there are associations between quality of life and treatment outcome (re-treatment rates or amount of pain relief). Measured on a continuous scale and will be compared between groups using 2-sample t-tests. Either multiple logistic regression (for binary outcomes) models or analysis of covariance (ANCOVA) models for continuous outcomes will be used. The QLQ-C15-PAL has high sensitivity and specificity for identifying clinically important symptoms and functional health impairments. Scores range from 0 to 100 with higher values indicating a better quality of life in the Physical and Emotional Functioning and Quality of Life categories. Higher scores in Symptoms Scales categories indicates a worse quality of life. Most questions are rated on a 4-point Likert scale (1 = not at all to 4 = very much), but the global quality of life item uses a 7-point scale (1 = very poor to 7 = excellent)
Time Frame: At 3 months and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 19 | 24
score on a scale
  Physical Functioning - 6 months | 87.0 (14.9) | 64.2 (31.3)
  Physical Functioning - 3 months | 65.7 (28.5) | 72.2 (24.9)
  Emotional Functioning - 3 months | 74.0 (30.5) | 75.4 (26.5)
  Emotional Functioning - 6 months | 84.7 (20.7) | 79.6 (27.1)
  Symptom Scales (3 months) - Dyspnea | 26.4 (29.5) | 22.7 (34.7)
  Symptom Scales (3 months) - Pain | 52.7 (30.3) | 52.2 (31.5)
  Symptom Scales (3 months) - Insomnia | 33.3 (31.1) | 27.3 (28.4)
  Symptom Scales (3 months) - Fatigue | 50.0 (30.0) | 47.8 (24.8)
  Symptom Scales (3 months) - Appetite loss | 37.5 (37.2) | 25.8 (25.1)
  Symptom Scales (3 months) - Nausea/vomiting | 22.2 (23.4) | 16.7 (19.9)
  Symptom Scales (3 months) - Constipation | 29.3 (30.9) | 31.9 (38.2)
  Quality of Life - 3 months | 62.7 (27.8) | 60.1 (24.5)
  Symptom Scales (6 months) - Dyspnea | 19.4 (26.4) | 31.5 (38.7)
  Symptom Scales (6 months) - Pain | 37.5 (28.5) | 55.6 (37.0)
  Symptom Scales (6 months) - Insomnia | 27.8 (34.3) | 40.7 (38.9)
  Symptom Scales (6 months) - Fatigue | 31.9 (26.1) | 48.1 (31.3)
  Symptom Scales (6 months) - Appetite loss | 25.0 (35.2) | 27.8 (38.3)
  Symptom Scales (6 months) Nausea/vomiting | 22.2 (21.7) | 33.3 (34.3)
  Symptom Scales (6 months) - Constipation | 16.7 (22.5) | 33.3 (28.0)
  Quality of Life - 6 months | 79.2 (12.6) | 63.9 (30.9)
Statistical Analysis 1: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Physical Functioning p-value at 3 months; Test type: Superiority; p = 0.4182, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Emotional functioning p-value at 3 months; Test type: Superiority; p = 0.8700, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Dyspnea at 3 months; Test type: Superiority; p = 0.7008, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scale Pain at 3 months; Test type: Superiority; p = 0.9562, t-test, 2 sided
Statistical Analysis 5: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scale Insomnia at 3 months; Test type: Superiority; p = 0.4951, t-test, 2 sided
Statistical Analysis 6: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scale Fatigue at 3 months; Test type: Superiority; p = 0.7868, t-test, 2 sided
Statistical Analysis 7: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scale Appetite loss at 3 months; Test type: Superiority; p = 0.2200, t-test, 2 sided
Statistical Analysis 8: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scale Nausea/vomiting at 3 months; Test type: Superiority; p = 0.7998, t-test, 2 sided
Statistical Analysis 9: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scale Constipation at 3 months; Test type: Superiority; p = 0.7998, t-test, 2 sided
Statistical Analysis 10: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scale Quality of Life at 3 months; Test type: Superiority; p = 0.7409, t-test, 2 sided
Statistical Analysis 11: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Physical Functioning at 6 months; Test type: Superiority; p = 0.0128, t-test, 2 sided
Statistical Analysis 12: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Emotional Functioning at 6 months; Test type: Superiority; p = 0.5861, t-test, 2 sided
Statistical Analysis 13: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Dyspnea at 6 months; Test type: Superiority; p = 0.3561, t-test, 2 sided
Statistical Analysis 14: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Pain at 6 months; Test type: Superiority; p = 0.1647, t-test, 2 sided
Statistical Analysis 15: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Insomnia at 6 months; Test type: Superiority; p = 0.3571, t-test, 2 sided
Statistical Analysis 16: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Fatigue at 6 months; Test type: Superiority; p = 0.1494, t-test, 2 sided
Statistical Analysis 17: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Appetite loss at 6 months; Test type: Superiority; p = 0.8424, t-test, 2 sided
Statistical Analysis 18: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Nausea/vomiting at 6 months; Test type: Superiority; p = 0.3287, t-test, 2 sided
Statistical Analysis 19: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Symptom Scales - Constipation at 6 months; Test type: Superiority; p = 0.0961, t-test, 2 sided

5. Secondary Outcome: Incidence of Adverse Events - Grade 3 or Higher
Description: Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Groups will be compared to determine whether there are any differences in the number or severity of toxicities. When comparing severity of toxicities between groups, chi-square tests will be examined. The Cochran-Armitage trend test can be used to determine if there is evidence a trend in severity of toxicities when comparing groups. Because of the patient population as well as the treatment, emphasis will be placed on gastrointestinal (GI disturbance, esophagitis, diarrhea, nausea, and vomiting), hematological (low blood counts or bleeding), spinal (bone fracture, compression fracture, insufficiency, or myelitis), and pulmonary toxicities (pneumonitis) and recorded by clinical research coordinators. Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to the event.
Time Frame: Up to 6 months post-treatment
Measure: Number; unit: participants
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 19 | 24
participants
  Nausea - Grade 3 | 1 | 0
  Nausea - Grade 4 | 0 | 0
  Nausea - Grade 5 | 0 | 0
  Anemia - Grade 3 | 0 | 1
  Anemia - Grade 4 | 0 | 0
  Anemia - Grade 5 | 0 | 0
  Diarrhea - Grade 3 | 0 | 1
  Diarrhea - Grade 4 | 0 | 0
  Diarrhea - Grade 5 | 0 | 0
  Fatigue - Grade 3 | 0 | 1
  Fatigue - Grade 4 | 0 | 0
  Fatigue - Grade 5 | 0 | 0
  Pain - Grade 3 | 0 | 1
  Pain - Grade 4 | 0 | 0
  Pain - Grade 5 | 0 | 0
  Dehydration - Grade 3 | 1 | 0
  Dehydration - Grade 4 | 0 | 0
  Dehydration - Grade 5 | 0 | 0
  Dyspnea - Grade 3 | 0 | 1
  Dyspnea - Grade 4 | 0 | 0
  Dyspnea - Grade 5 | 0 | 0

6. Secondary Outcome: Participants With Patient Satisfaction of Treatment Outcome - Patient Satisfaction With Cancer Care (PSCC-18)
Description: Analyses will be performed that examine whether there are associations between patient satisfaction and treatment outcome (re-treatment rates or amount of pain relief). Satisfaction will be measured by answering a series of questions with a scoring scale range of 1 (strongly agree) to 5 (strongly disagree). The scoring range for the Patient Satisfaction with Cancer Care (PSCC)-18 is 18 (best score) to 90 (worse score). A lower total score indicates higher satisfaction with cancer care.
Time Frame: At 3 months and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 19 | 24
score on a scale
  3 months | 25.8 (8.9) | 26.3 (8.2)
  6 months | 25.4 (10.0) | 26.0 (10.1)
Statistical Analysis 1: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; At 3 months, total score for PSCC-18; Test type: Superiority; p = 0.8444, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; At 6 months, total score for PSCC-18; Test type: Superiority; p = 0.8946, t-test, 2 sided

7. Secondary Outcome: Participants With Perceived Stress of Treatment Outcome - Perceived Stress Scale (PSS-10)
Description: The Perceived Stress Scale (PSS) is a stress assessment instrumentto help understand how different situations affect feelings and perceived stress. Scoring scale is 1 (never) to 4 (very often) when monitoring stress, the higher the total score the more stress the participant has experienced. The Perceived Stress Scale (PSS-10) is scored by summing the responses to all 10 items, with a total score ranging from 0 to 40. To get the score, you first need to reverse the scoring for the positively worded items (items 4, 5, 7, and 8). A total score of 0-13 suggests low stress, 14-26 indicates moderate stress, and 27-40 represents high stress.
  Perceived helplessness (items 1, 2, 3, 6, 9, 10) - measuring an individual's feelings of a lack of control over their circumstances or their own emotions or reactions.
  Lack of self-efficacy (items 4, 5, 7, 8) - measuring an individual's perceived inability to handle problems.
Time Frame: At 3 months and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 19 | 24
score on a scale
  Perceived helplessness total (3 months) | 8.7 (5.6) | 8.0 (6.1)
  Perceived self-efficacy total (3 months) | 5.6 (3.6) | 4.7 (3.7)
  Total PSS-10 score (3 months) | 14.2 (8.1) | 13.0 (8.6)
  Perceived helplessness total (6 months) | 5.9 (4.4) | 8.6 (6.9)
  Perceived self-efficacy total (6 months) | 4.7 (3.4) | 5.6 (4.4)
  Total PSS-10 score (6 months) | 10.6 (7.2) | 14.5 (10.7)
Statistical Analysis 1: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Perceived helplessness total at 3 months; Test type: Superiority; p = 0.6700, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Perceived self-efficacy total at 3 months; Test type: Superiority; p = 0.4350, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Total PSS-10 score at 3 months; Test type: Superiority; p = 0.6131, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Perceived helplessness total at 6 months; Test type: Superiority; p = 0.2518, t-test, 2 sided
Statistical Analysis 5: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Perceived self-efficacy total; Test type: Superiority; p = 0.5529, t-test, 2 sided
Statistical Analysis 6: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Total PSS-10 score at 6 months; Test type: Superiority; p = 0.2833, t-test, 2 sided

8. Secondary Outcome: Participants With Social Support Assessed Via Self-Reported Surveys
Description: Association between social support and treatment outcomes will be assessed. Social support will be measured by answering a series of questions with a scoring scale range of 1 (definitely false for you) to 4 (definitely true for you). The total score is the sum of all items, ranging from 0 to 36. Sum the scores for the four items in each subscale (Appraisal, Belonging, and Tangible) to get a score ranging from 0 to 12 for each subscale. The higher the total score the more support the participants receive from their support network.
Time Frame: At 3 months and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Control) 8 Gy x 1 | Arm B (Treatment) 8 Gy x 2
Number analyzed (Participants) | 19 | 24
score on a scale
  Appraisal Support subscale total (3 months) | 6.5 (1.5) | 6.0 (1.7)
  Belonging Support subscale total (3 months) | 5.8 (1.4) | 6.0 (1.9)
  Tangible Support subscale total (3 months) | 8.1 (1.7) | 8.8 (1.7)
  Total ISEL score (3 months) | 20.2 (3.3) | 20.8 (4.3)
  Appraisal Support subscale total (6 months) | 6.3 (1.3) | 6.1 (0.8)
  Belonging Support subscale total (6 months) | 6.2 (2.0) | 6.6 (1.1)
  Tangible Support subscale total (6 months) | 8.5 (1.4) | 8.7 (1.0)
  Total ISEL score (6 months) | 20.9 (2.2) | 21.4 (1.4)
Statistical Analysis 1: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Appraisal Support subscale total at 3 months; Test type: Superiority; p = 0.3784, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Belonging Support subscale total at 3 months; Test type: Superiority; p = 0.6640, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Tangible Support subscale total at 3 months; Test type: Superiority; p = 0.1745, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Total ISEL score at 3 months; Test type: Superiority; p = 0.5792, t-test, 2 sided
Statistical Analysis 5: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Appraisal Support subscale total at 6 months; Test type: Superiority; p = 0.6814, t-test, 2 sided
Statistical Analysis 6: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Belonging Support subscale total at 6 months; Test type: Superiority; p = 0.5219, t-test, 2 sided
Statistical Analysis 7: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Tangible Support subscale total; Test type: Superiority; p = 0.5516, t-test, 2 sided
Statistical Analysis 8: Comparison: Arm A (Control) 8 Gy x 1 vs Arm B (Treatment) 8 Gy x 2; Total ISEL score at 6 months; Test type: Superiority; p = 0.4329, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 6 months post-treatment, 6 months in Arm I (8 Gy x 1 fraction) and 6 months and 1 week for Arm II (8 Gy x 2 fractions)
Arm/Group | ARM I (Palliative Radiation Therapy) | ARM II (Palliative Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 19/51 | 17/51
Serious Adverse Events (participants affected / at risk) | 19/51 | 37/51
Other Adverse Events (participants affected / at risk) | 32/51 | 32/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM I (Palliative Radiation Therapy) (N=51) | ARM II (Palliative Radiation Therapy) (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Death, NOS (General disorders) | 19 (19) | 17 (17)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury, poisoning and procedures complications, other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney pain (Renal and urinary disorders) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM I (Palliative Radiation Therapy) (N=51) | ARM II (Palliative Radiation Therapy) (N=51)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 7 (8)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (6)
Chills (General disorders) | 0 (0) | 1 (1)
Edema, limbs (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 4 (4) | 10 (10)
Fever (General disorders) | 1 (1) | 1 (2)
Non-cardiac chest pain (General disorders) | 5 (5) | 3 (3)
Pain (General disorders) | 7 (8) | 12 (12)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestation (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (3)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Weight loss (Investigations) | 4 (4) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT02699697/Prot_SAP_001.pdf
  • Informed Consent Form (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT02699697/ICF_000.pdf